CLINICAL TRIAL: NCT00580515
Title: Randomized Controlled Trial of Family Focused Grief Therapy in Palliative Care and Bereavement
Brief Title: Trial of Family Focused Grief Therapy in Palliative Care and Bereavement
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Beth Israel Medical Center (Other); Calvary Hospital, Bronx, NY (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 05-120; CA115329
Record Dates: First submitted 2007-12-20; First posted 2007-12-24 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: Cancer; Randomized Controlled Trial; Family Therapy intervention
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

ARMS (3):
- 1 (Experimental): 6 sessions of Family Focused Group Therapy
  Interventions: Behavioral: Family Focused Group Therapy
- 2 (Experimental): 10 Sessions of Family Focused Group Therapy
  Interventions: Behavioral: Family Focused Group Therapy
- 3 (Active Comparator): Standard Care- Social work consultations are routinely provided to the cancer patients, but relatives are only seen during admissions or upon request
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Family Focused Group Therapy — 6 Sessions of Family Focused Group Therapy (FFGT). The FFGT intervention will have assessment, focused therapy, consolidation, and termination phases. The first two sessions are assessment sessions and occur one week apart. There will be two or six focused intervention sessions depending on the predetermined length of therapy. The first focused intervention session is approximately two weeks after the last assessment session. Subsequent focused intervention sessions are expected to follow once every month. Finally, there will be two consolidation/termination sessions, which will occur one time each, approximately two months apart. The six session program is expected to extend over a period of 6 months and the 10 session program over 10 months.
  Other Names: FFGT
  Arms: 1; 2
Behavioral: Family Focused Group Therapy — 10 Sessions of Family Focused Group Therapy (FFGT). The FFGT intervention will have assessment, focused therapy, consolidation, and termination phases. The first two sessions are assessment sessions and occur one week apart. There will be two or six focused intervention sessions depending on the predetermined length of therapy. The first focused intervention session is approximately two weeks after the last assessment session. Subsequent focused intervention sessions are expected to follow once every month. Finally, there will be two consolidation/termination sessions, which will occur one time each, approximately two months apart. The six session program is expected to extend over a period of 6 months and the 10 session program over 10 months
  Other Names: FFGT
  Arms: 1; 2
Behavioral: Standard of Care — Standard of Care Families assigned to the Usual Care Condition will receive standard psychosocial care which is based on the following patterns: Social work consultations are routinely provided to the cancer patients, but relatives are only seen during admissions or upon request.
  Arms: 3

SUMMARY:
The purpose of this study is to learn how well family therapy works if given while a family member is being treated for a serious illness and whether it helps their family to continue meeting for a time after their death. The therapy aims to assist the family communication and support during both palliative care and bereavement. The investigators also want to learn how many family therapy sessions spread out over time are best for helping patients and their families.

Patients are randomly assigned to one of three groups: patients who receive standard palliative care, patients and their families who take part in 6 sessions, and patients and their families who take part in 10 sessions.

DETAILED DESCRIPTION:
This Randomized Controlled Trial (RCT) seeks to test the efficacy and dose responsiveness of a manualized family therapy intervention called Family Focused Grief Therapy (FFGT), which is delivered to families of patients with advanced disease and continued into bereavement. Randomization is to three arms: 6 sessions of FFGT, 10 sessions of FFGT, or standard care. The study also explores the potential mediators of effective outcome, empowering further refinement of the intervention, and undertakes an analysis of health-related costs of bereavement care. It is a multi-site study involving Memorial Hospital for Cancer and Allied Diseases (a comprehensive cancer center), Calvary Hospital (a dedicated palliative care hospital with home hospice care program)and Beth Israel (a medical center with a dedicated pain and palliative care department. Consenting families will be assessed at baseline through completion of questionnaires that appraise each individual's psychosocial well-being and perception of their family's functioning. Therapy will be delivered by family therapists (social workers, psychologists, and psychiatrists), who will attend regular supervision sessions to sustain fidelity of the model of intervention. Follow-up of family members for psychosocial well-being, perceptions of family functioning, and costs of heath-related care will occur at 3, 6, 9, & 13 months after the patient's death or completion of therapy sessions.

ELIGIBILITY:
Inclusion Criteria:

Subject/Patient Inclusion Criteria

* Individuals with advanced disease/Stage 4-IV cancer who may be involved in palliative care treatment program.
* Individuals with a poor prognosis Patient and Family Member Inclusion Criteria.
* Per investigator's judgment participants must have satisfactory cognitive functioning to provide valid informed consent and participate in family therapy.
* In the event that the index family member is declining or too frail to take part in family meetings, the family is able to participate without the index patient being involved in the study.
* For every enrolled family there must be at least 2 family members willing/able to take part at the time of recruitment.
* The presence of FRI screening scores of ≤ 9 or cohesiveness subscale score < 4 based on the perception of any single family member, including the patient.

Exclusion Criteria:

* Inability through language to complete the study questionnaires - inability to speak English with an English-speaking therapist.
* Age less than 12 years old for a child.
* Patient and family member determined geographical inaccessibility to attend family sessions.
* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude participation in a psychotherapeutic intervention.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2005-11; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy and dose responsiveness of family intervention in preventing bereavement and depression compared with standard palliative care among family members and to examine whether distress moderates impact of FFGT | 5 years

SECONDARY OUTCOMES:
Evaluate whether family coping and communication mediate the impact of FFGT and examine costs of FFGT and standard palliative care, and whether the additional costs are offset by reductions in community health utilization | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Talia Zaider, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Beth Israel Hospice Program, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Calvary Hospital, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan-Kettering web site — http://www.mskcc.org